CLINICAL TRIAL: NCT03630107
Title: In-Use Test of a Shampoo (WO 5101) in Subjects With Pruritus of the Scalp
Brief Title: In-Use Test of a Cosmetic Product in Subjects With Chronically Itchy Scalp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: SIT Skin Investigation and Technology Hamburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS-05/2017
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Pruritus of the Scalp
Keywords: itchy scalp; chronic pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WO 5101 Shampoo for Scalp and Hair (Experimental): WO 5101 is used in subjects with chronically itchy scalp
  Interventions: Other: WO 5101 Shampoo for Scalp and Hair

INTERVENTIONS:
Other: WO 5101 Shampoo for Scalp and Hair — Wash the hair at least three times a week for a period of four weeks

SUMMARY:
The aim of the study is to evaluate the tolerance of the Shampoo (WO 5101) on the scalp by a dermatologist and by the subjects themselves after four weeks of regular product use.

Additional objective of this clinical in-use study was to evaluate the cosmetic features and the acceptance of the product by means of a questionnaire at the end of the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* age: ≥ 18 years
* with chronically itchy scalp
* normal to dry scalp or scalp prone to neurodermatitis

Exclusion Criteria:

* any deviation from the above-mentioned criteria
* users of sour hair conditioner
* subjects who wash their hair more than once a day
* other dermatological disorders (scars, moles) on the scalp
* known incompatibilities to cosmetics and ingredients of cosmetic test products (please see INCI)
* topical medication in the test area within 1 month prior to study start
* systemic medication with anti-inflammatory agents and antibiotics within two weeks prior to starting of the study
* systemic medication with retinoids, antihistamines and/or immunomodulators (e.g. cortisone, corticosterone, chemotherapeutic agents) within four weeks prior to starting of the study
* severe internistic disease that leads to pruritus

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Dermatological Tolerance of the Test Product on the Scalp | baseline, four weeks
  Change from Baseline at four weeks by the means of a dermatological assessment of scalp
  1. erythema
  2. edema
  3. dryness
  4. scaliness
  5. papules
  6. pustules
  7. fissures
  8. pruritus
  9. burning
  10. Tension
  all Parameters (a-j) were assessed by 6-tiered rating scale with 0.5 intervals (0=absent; 0.5=very slight, 1/1.5= slight; 2/2.5=moderate; 3/3.5=severe and 4=extreme)
Subjective Tolerance of the Test Product on the Scalp | baseline, four weeks
  Change from baseline at four weeks by means of a self-assessment questionnaire (with 13 questions regarding cosmetic features of the product as well as satisfaction with cosmetic performance).

SECONDARY OUTCOMES:
Cosmetic Features of the Test Product | baseline, four weeks
  Change from Baseline for the Cosmetic Features (scalp feeling after application, fragrance, hair styling, combability, lightness of the hair) of the Test Product by the means of a questionnaire
Reduction of Pruritus | baseline, four weeks
  Change from Baseline Reduction of Pruritus at four weeks by the means of a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Söhl, MD, Study Director — Dermatologist
Locations (1):
- SIT Skin Investigation and Technology Hamburg GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No